CLINICAL TRIAL: NCT02393664
Title: Effects of Nonintubated Versus Intubated General Anesthesia on Recovery After Thoracoscopic Lung Resection: A Prospective Randomized Trial
Brief Title: Effects of Nonintubated Versus Intubated General Anesthesia on Recovery After Thoracoscopic Lung Resection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201410045RINB
Record Dates: First submitted 2015-03-08; First posted 2015-03-19 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Lung Neoplasms
Keywords: Thoracoscopy; Recovery; Tracheal intubation
MeSH Terms: conditions — Lung Neoplasms | interventions — Propofol; Bupivacaine; Sevoflurane; Rocuronium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nonintubated group (Experimental): Patients undergoing thoracoscopic surgery using nonintubated technique with propofol and bupivacaine.
  Interventions: Drug: propofol, bupivacaine
- Intubated group (Active Comparator): Patients undergoing thoracoscopic surgery using intubated general anesthesia with sevoflurane and rocuronium.
  Interventions: Drug: sevoflurane, rocuronium

INTERVENTIONS:
Drug: propofol, bupivacaine — Nonintubated technique for thoracoscopic surgery using propofol infusion, intercostal and vagal blocks with bupivacaine infiltrations.
  Other Names: Fresofol, Marcaine
  Arms: Nonintubated group
Drug: sevoflurane, rocuronium — Conventional intubated general anesthesia for thoracoscopic surgery using sevoflurane and rocuronium, and tracheal intubation with a double-lumen tube or a endobronchial blocker.
  Other Names: Ultane, Esmeron
  Arms: Intubated group

SUMMARY:
Lung cancer is the leading cause of cancer death in Taiwan and worldwide. With the advancement of thoracoscopic technique, thoracoscopic surgery has emerged as a reasonable option for the management of early-stage non-small cell lung cancer (NSCLC). Additionally, current lung cancer screening policy recruits increasing number of candidates requiring thoracoscopic lung resections because of lung nodules/tumors. Traditionally, intubated general anesthesia with one-lung ventilation using a double-lumen endotracheal tube or an endobronchial blocker has been considered mandatory in thoracoscopic surgery. However, adverse effects of intubated general anesthesia are not negligible. Recently, a nonintubated thoracoscopic technique has developed to reduce the adverse effects of intubated general anesthesia with encouraging results. Nonetheless, the role of nonintubated technique in thoracoscopic lung resection surgery in quality of postoperative recovery in not clear. As an enhanced recovery is the major goal of modern minimally invasive surgery, the investigators hypothesize that nonintubated thoracoscopic technique can facilitate and improve the recovery quality after surgery. To this end, the investigators will recruit 300 patients in subgroups including patients undergoing segmentectomy/lobectomy, wedge resection and geriatric patients in this two-year project. Patients will be randomly allocated in nonintubated and intubated groups and quality of recovery of all patients will be evaluated according the protocol of Postoperative Quality of Recovery Scale. In the meantime, the preoperative and postoperative cytokines will be compared between the groups as well as patients with different recovery scales.

DETAILED DESCRIPTION:
Treatment protocol of nonintubated technique and intubated general anesthesia

Nonintubated technique: All nonintubated patients will be premedicated with 50 to 100 μg of fentanyl intravenously and will be continuously monitored electrocardiographically, along with pulse oximetry, respiratory rate, blood pressure, body temperature, and urine output. End-tidal carbon dioxide will be continuously monitored by insertion of a detector into one nostril. A bispectral index sensor (BIS Quatro, Aspect Medical System, Norwood, MA, USA) will be applied to the forehead of each patient to monitor the level of consciousness. Additionally, a non-invasive near-infrared cerebral regional oximetry (INVOSTM 5100BINVOS 5100B Cerebral Oximeter, Somanetics Corporation, Troy, MI, USA) will be applied to monitor the regional oxygen saturation of the brains. The patients will be sedated with intravenous propofol (Fresol 1%, Fresenius Kabi GmbH, Graz, Austria) using a target-controlled infusion method (Injectomat® TIVA Agilia, Fresenius Kabi GmbH, Graz, Austria). The level of sedation will be set to achieve a bispectral index value between 40 and 60, and incremental intravenous injections of fentanyl 25 μg will be given to maintain a respiratory rate between 12 and 20 breaths/min. Oxygen will be supplied through a ventilation mask.

Conventional intubated general anesthesia: All intubated patients will be monitored as for nonintubated patients. Anesthesia will be induced by intravenous administration of propofol (1 - 2.5 mg/kg), fentanyl (100 μg), and rocuronium (0.6 mg/kg) and will be maintained by sevoflurane and rocuronium at the discretion of anesthesiologist and bispectral index monitoring. A double-lumen endotracheal tube or endobronchial blocker will be inserted for one lung isolation during the procedure and a bronchoscopy will be used to facilitate the correct isolation of targeted bronchus at the discretion of anesthesiologist. The dependent lung will be ventilated using protective lung strategy with a tidal volume of 6 to 8 mL/kg, a respiratory rate of 10 to 16 breaths/min to maintain the arterial carbon dioxide tension at 35 to 45 mmHg. After the operation, the patients will be extubated in the operating room or remain intubated and be sent to the intensive care unit at the discretion of anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Age: older than 20 years old;
* Tumor size less than 6 cm;
* Eligible for unilateral thoracoscopic surgery;
* Preoperative lung function FEV1 > 60%.

Exclusion Criteria:

* Neurological deficits, including previous stroke, dementia etc.;
* Previous thoracic surgery;
* Suspect invasion of tumor into chest wall, diaphragm, or main bronchus;
* Suspect severe pleural or diaphragmatic adhesions;
* Significant comorbidities with high ASA classification (ASA > 3), including history of heart failure, liver failure and renal failure;
* Severe obstructive sleep apnea requiring continuous positive airway pressure support or oxygen supplement;
* Difficult airway management;
* Pregnant women.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative Quality of Recovery Scale (PQRS) | 1 month
  PQRS is a measure tool to evaluate the patient recovery after surgery, which includes five domains, i.e., physiological factors, nociceptive factors, emotional factors, recovery of activity of daily life and cognitive factors.

SECONDARY OUTCOMES:
Composite outcomes, including perioperative adverse effects, mortality, ICU stay, hospital stay, ventilator use, etc. | 1 month
Changes of inflammatory cytokines before and after surgery. | 3 days
  Inflammatory responses

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shing Chen, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan